CLINICAL TRIAL: NCT05621291
Title: A Pilot Trial to Evaluate Next-Generation Sequencing (NGS) Testing and Monitoring of B-Cell Recovery to Guide Management Following CAR T-cell Induced Remission in Pediatric Patients With B Lineage Acute Lymphoblastic Leukemia
Brief Title: A Study to Evaluate Next-Generation Sequencing (NGS) Testing and Monitoring of B-cell Recovery to Guide Management Following Chimeric Antigen Receptor T-cell (CART) Induced Remission in Children and Young Adults With B Lineage Acute Lymphoblastic Leu...
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000792; 000792-C
Record Dates: First submitted 2022-11-16; First posted 2022-11-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-11

CONDITIONS: B-All; Acute Lymphoblastic Leukemia
Keywords: B-All; Car-Cure; Result Monitoring
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/Intervention (Experimental): Systematic, frequent monitoring intervention to risk stratify pts for risk of relapse postCART
  Interventions: Diagnostic Test: NGS testing

INTERVENTIONS:
Diagnostic Test: NGS testing — antigen immunophenotype agnostic approach for disease detection using blood and bone marrow samples

SUMMARY:
Background:

Chimeric antigen receptor T-cell (CART) therapy is a form of immunotherapy which can be used to treat people with relapsed B-ALL. For those who achieve remission after CART alone, it may cure up to 50% of people who receive this therapy. However, for people who relapse after CART, it can be hard to achieve remission again. In patients where CART fails, stem cell transplant (HCT) can be used to prevent relapse and achieve cure. But HCT can cause serious side effects. Better testing is needed to distinguish people who can be cured with CART alone from people who may also need to have HCT.

Objective:

To see if the use of a series of blood and bone marrow tests at regular intervals can help monitor for B-ALL relapse after CART therapy.

Eligibility:

People aged 1 to 25 years with B-ALL who have had CART therapy within the past 42 days. They must never have had a blood stem cell transplant; they must also have no measurable blood cancer cells.

Design:

Participants will visit the clinic every 2 weeks starting 42 days after they receive CART therapy. Each visit will be about the same amount of time as a regular clinic visit. about 8 hours.

Participants will have blood drawn for testing on each visit.

Bone marrow biopsy/aspirate will be done during 4 of the visits at routine timepoints after CART. A needle will be inserted to draw a sample of tissue from inside the bone in the hip.

A small amount of blood and tissue will be tested with ClonoSEQ and to evaluate for normal B-cells side by side with the standard tests.

The combined testing may help determine whether participants are eligible for HCT and/or at risk of relapse after CART.

Participants will be in the study for 2 years.

DETAILED DESCRIPTION:
Background:

* Given the dismal outcomes for patients who experience a relapse following CD19 CART and the potential for using Hematopoietic cell transplantation (HCT) for post-CART remission consolidation for relapse prevention, there is a clear opportunity to improve outcomes for patients with B-ALL who proceed to CART. With a goal of improving overall survival, it remains critically important to be able to predict which patients are at high risk of relapse in whom an HCT would be indicated for remission consolidation. Distinguishing this high-risk cohort from low-risk patients who are able to maintain durable remission following CART and in whom HCT-associated toxicities could be avoided is equally important.
* Thus, in the context of this biomarker-based study, we propose a systematic approach utilizing the best-known biomarkers for remission monitoring which assess both functional CART persistence and incorporates antigen immunophenotype agnostic approach for disease detection will improve LFS post CD19 CART.

Objective:

-To assess efficacy of a novel biomarker-guided risk-based strategy to monitor remission, both by assessing functional CART persistence and incorporating antigen immunophenotype agnostic approach (NGS monitoring) for disease detection, to inform decisions regarding post-CART HCT needed intervention, and to successfully collect biomarker samples at the scheduled times in enrolled HCT naive B-ALL participants receiving CD19 CART.

Eligibility:

* Age >=1 year and <= 25 years old at the time of CD19 CART infusion
* Diagnosis of CD19+ B-ALL in a bone marrow morphologic complete remission and are flow cytometry measurable residual disease (MRD) negative within 42 days post CD19 CART infusion.
* Must have an allogeneic HCT donor identified for potential HCT
* B-cell aplasia post CD19 CART persisting until the time of the first on-study intervention

Design:

-This single-arm multicenter study will enroll pediatric and young adult participants to evaluate the feasibility, and potential efficacy, of a risk-based, biomarker-driven, consolidation HCT strategy following CD19 CART.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >=1 year and <= 25 years old at the time of CD19 CART infusion
* Confirmed diagnosis of CD19+ B-ALL with an informative NGS clonality sample

  --Have an informative NGS clonality sample for MRD assessment based on immunoglobulin rearrangement in bone marrow or blood at any time of active disease between diagnosis and CD19 CART infusion and any time prior to the first on-study intervention confirmed by NGS MRD testing.
* Post-CD19 CART infusion disease status:

  * Are in bone marrow morphologic complete remission and are flow cytometry measurable residual disease (MRD) negative within 42 days post CD19 CART infusion.
  * Are NGS MRD negative by tracking sample in the bone marrow within 42 days post CD19 CART infusion confirmed by NGS MRD testing.
* Received first CD19 (4-1BB) CART within 42 days prior to enrollment. Note: Eligible CART including FDA approved Kymriah (tisagenlecleucel) infused on a treatment plan, research study, or other comparable 4-1BB based constructs.

Study chairs will determine whether other 4-1BB CART are considered comparable.

* All participants must have an allogeneic HCT donor identified for potential HCT. Note: Donor identification and selection will be according to institutional practice.
* Have B-cell aplasia (BCA) post CD19 CART persisting within 42 days post CD19 CART infusion. Note: BCA persisting is defined as <1% B cells lymphocytes or <50 B cells/microliter in the peripheral blood
* Performance of all screening tests prior to day 42 post CD19 CART.
* The ability of participant or parent/guardian to understand and the willingness to sign a written consent document or participants unable to consent if they are represented by a Legally Authorized Representative (LAR).

EXCLUSION CRITERIA:

* Prior hematopoietic stem cell transplantation (HCT)
* Recent history of the extramedullary disease (EMD) that requires ongoing radiographic surveillance (e.g., participants with active EMD at CD19 CART infusion that requires monitoring by imaging without the ability to more precisely assess disease status will be ineligible). A remote history of EMD does not exclude the participant.
* Active and/or residual central nervous system (CNS) disease that requires ongoing therapy or monitoring.
* Co-morbidities precluding myeloablative HCT. Note: Determination of co-morbidities precluding myeloablative HCT will be made by the treating transplant (HCT) physician and documented in the research record. This does not require that the participant is immediately fully eligible for HCT, only that there are no long-term comorbidities that would preclude a myeloablative approach (e.g., renal failure, severe cardiac failure, long-term oxygen requirement).
* Uncontrolled, symptomatic, intercurrent illness or social situations that would limit compliance with study requirements. Note: Determination of uncontrolled, symptomatic illness or social situation that would limit compliance with the study requirements will be made by the site-PI and documented in the research record.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of novel biomarker-guided risk based strategy to monitor remission | baseline to 1 year post CD19 CART infusion
  NGS MRD testing of blood and bone marrow samples and evaluation of BCA

SECONDARY OUTCOMES:
Time to relapse | baseline to 1 year post CD19 CART infusion
  Defined as time from CART cell infusion to relapse
Time to HCT | baseline to 1 year post CD19 CART infusion
  Defined as time from CART cell infusion to receiving HCT
Leukemia Free Survival | baseline to 1 year post CD19 CART infusion
  Defined as time from CART cell infusion to first occurrence of relapse or death
Overall survival | baseline to 1 year post CD19 CART infusion
  Defined as time from CART cell infusion to death

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (8):
- United States (8):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber/Boston Children s Hospital, Boston, Massachusetts
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Seattle Children's, University of Washington, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be made available within 10 years after completion of the primary endpoint. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000792-C.html